CLINICAL TRIAL: NCT01635374
Title: Per-Oral Endoscopic Esophagomyotomy (POEM)
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Eric Hungness, Assistant Professor of Surgery, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU00030841
Record Dates: First submitted 2012-04-10; First posted 2012-07-09 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Per-Oral Endoscopic Esophagomyotomy (Experimental): Patients will have a standard pre-operative work-up that may include upper endoscopy (EGD), endoscopic ultrasound (EUS), upper GI X-rays, high-resolution manometry, pH, FLIP and impedance measurement studies. Once a diagnosis of esophageal motility disorder is confirmed, patients will be offered POEM or standard treatment. Patients undergoing POEM will review and sign the study consent prior to their procedure. Patients will return and be evaluated two weeks following their procedure. At this visit, any post-operative complications will be noted in the patient's medical record. Also, at this visit and at the preoperative visit, patients will complete a standardized Quality of Life assessment. Perceived pain levels and type and frequency of pain medications will be recorded in the patient's medical record. Patients will then return at 6 weeks post-op to complete a second set of questionnaires and have a high resolution manometry performed to assess residual LES pressure.
  Interventions: Procedure: Per-Oral Endoscopic Esophagomyotomy

INTERVENTIONS:
Procedure: Per-Oral Endoscopic Esophagomyotomy — In this procedure, performed in the operating room under general anesthesia, a flexible endoscope is passed into the esophagus, a mucosal flap and a submucosal tunnel is created. This tunnel extends onto the stomach. The inner circular muscle layer of the lower esophagus and sphincter (LES) is identified and a myotomy is started 3-4cm distal to the mucosal flap and carried all the way onto the stomach. The mucosal opening is then closed with standard endoscopic clips. Patients will be admitted to the hospital and a gastrograffin esophagram will be performed on post-op day 2 to rule out esophageal leak. A standardized symptom checklist will be used to assess patient's prior to hospital discharge and on post-op days 4 and 7. All patient will have a 2 week post-op appointment.
  Other Names: POEM

SUMMARY:
Achalasia is an esophageal motility disease that usually requires surgical intervention (esophagomyotomy). Laparoscopic techniques have reduced the morbidity associated with myotomy, but post-op GERD, wound infection, hernia and incisional pain are common. A new NOTES based procedure, per-oral endoscopic esophagomyotomy (POEM), has been developed that eliminates the need for skin incisions. All patients enrolled in this study, will have a thorough pre-op workup (including upper endoscopy, upper GI radiographs, high resolution esophageal manometry) confirming the diagnosis of achalasis at the Northwestern Esophageal Center. In this procedure, performed in the operating room under general anesthesia, a flexible endoscope is passed into the esophagus, a mucosal flap and a submucosal tunnel is created. This tunnel extends onto the stomach. The inner circular muscle layer of the lower esophagus and sphincter (LES) is identified and a myotomy is started 3-4cm distal to the mucosal flap and carried all the way onto the stomach. The mucosal opening is then closed with standard endoscopic clips. Patients will be admitted to the hospital and a gastrograffin esophagram will be performed on post-op day 1 to rule out esophageal leak. All patient will have a 2-3 week post-op appointment

Patients with a confirmed diagnosis of achalasia may be offered POEM. The investigators hypothesize that POEM is feasible and safe and can effectively reduce residual LES pressure (as determined by manometry) and improve patients symptoms and quality of life.

DETAILED DESCRIPTION:
In this study, the investigators propose to use a surgical technique that eliminates skin incisions in patients undergoing esophagomyotomy. All patients will have a standard pre-operative esophageal work-up that may include upper endoscopy (EGD), endoscopic ultrasound (EUS), upper GI X-rays, high-resolution manometry, pH, FLIP and impedance measurement studies. Once the diagnosis of achalasia is confirmed, patients will be offered POEM or standard treatment for achalasia. All patients undergoing POEM will review and sign the study consent prior to their procedure.

Operative and recovery room times as well as hospital length of stay will be collected. During the hospital stay, severity of pain, use of pain medications and complications will be recorded. Patients will remain NPO for 1 day. Post-op day 1, all patient will receive an esophagram to rule out esophageal perforation. If normal, patients will be started on clear liquids and advanced to a full liquid diet for 1 week post-op.

Patients will return and be evaluated by their surgeon two weeks following their procedure. At this visit, any post-operative complications will be noted in the patient's medical record. Additionally at this visit and at the preoperative visit, patients will complete a standardized Quality of Life (QOL) assessment (i.e., SF-36). Perceived pain levels and type and frequency of pain medications will be recorded in the patient's medical record. Patients will then return at 6 weeks post-op to complete a second set of questionnaires and have a high resolution manometry performed to assess residual LES pressure.

The potential advantages to the patients entered into this study include those mentioned above regarding elimination of post-operative wound infection and hernia but also the lack of abdominal incisions may reduce pain and recovery time and likely have a cosmetic advantage as well. Potential risks of this study include those associated with use of flexible endoscopic instruments include esophageal perforation, bleeding and sore throat. In addition, there is the possibility that there may be new, unanticipated complications from this modified surgical technique. Patient risks will be mitigated by having the procedure performed by a surgeon with expertise in laparoscopic esophageal surgery, flexible endoscopy and NOTES, as well as having involvement of a skilled interventional gastroenterologist if deemed necessary. The principle investigator (who will be the primary surgeon for all procedures) has performed multiple pre-clinical animal and cadaver POEM procedures and has traveled to Yokohama, Japan to observe human POEM cases performed by Dr. Haru Inoue.

This feasibility study will initially evaluate the potential benefit, risks and impact on the patient's quality of life of this modified surgical technique in 20 patients. Once a standardized technique is established and risks are shown to be low, a prospective comparative evaluation is planned to compare this modified technique to the standard laparoscopic approach.

ELIGIBILITY:
Inclusion Criteria:

* Ability to undergo general anesthesia
* Age > 18 yrs. of age and < 85 yrs. of age
* Ability to give informed consent
* Confirmed diagnosis of achalsia, hypertensive lower esophageal sphincter, nutcracker esophagus, or diffuse esophageal spasm

Exclusion Criteria:

* Contraindicated for EGD
* Pregnancy
* Barrett esophagus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Change in Eckardt symptom score | inital pre-op surgical evaluation and one-year postoperative
  a brief 4 question survey will be filled out

SECONDARY OUTCOMES:
Number and frequency of intraoperative and postoperative complications | day of operation to one-year postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Eric S Hungness, M.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States